CLINICAL TRIAL: NCT06435078
Title: Developments of Novel Virtual Visual and Haptic Stimulation Systems for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Fong Chin Su, Chair Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B-ER-105-238
Record Dates: First submitted 2024-05-22; First posted 2024-05-30 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Healthy Elderly; Alzheimer Disease
Keywords: Pressing Evaluation and Training System; Virtual Reality; Augmented Reality
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR-mPETS (Experimental): subjects will be instructed to execute simulated piano playing tasks with Augmented Reality.
  Interventions: Device: mPETS(modified-PETS system)
- VR-mPETS (Active Comparator): subjects will be instructed to execute simulated piano playing tasks with Virtual Reality.
  Interventions: Device: mPETS(modified-PETS system)

INTERVENTIONS:
Device: mPETS(modified-PETS system) — The pressing evaluation and training system (PETS) consists of five force transducers, a pad position-adjustable frame, and biofeedback system. Five force transducers are used to collect the applied normal force from five digits.

SUMMARY:
previous studies indicated that sensory input can have positive impacts on finger force control in the elderly. Additionally, according to previous reports, apart from pharmacotherapy, nonpharmacologic interventions, such as psychosocial-environmental treatments, are emerging for the behavior and affective symptoms in AD . Moreover, enhanced finger force control and coordination lead to better hand dexterity and is believed to eventually improve life independence in the healthy elderly and the elderly with AD. Therefore, this study aims to develop novel virtual visual and haptic stimulation systems for the elderly to enhance their finger force control.

ELIGIBILITY:
Healthy elderly

Inclusion Criteria:

* Aged ≥ 65
* Healthy adult (no skeletal muscle, neurological disease that will affect training).

Exclusion Criteria:

* Neurological disorders
* Musculoskeletal problems
* History of surgery Patients with Alzheimer's disease

Inclusion Criteria:

* Diagnosed with Alzheimer's disease.
* No skeletal muscle, neurological disease that will affect training.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

PRIMARY OUTCOMES:
Force-track testing | Before and after intervention (4 weeks)
  Subjects will be asked to track the target force and presses task digit to fit the target line until finish.

SECONDARY OUTCOMES:
Sequential testing( reaction time) | Before and after intervention (4 weeks)
  In sequential testing, subjects will be asked to follow the pressing guide. The reaction time of sequential movements will be recorded and calculated.
Sequential testing( correct ratio ) | Before and after intervention (4 weeks)
  In sequential testing, subjects will be asked to follow the pressing guide. The correct ratio of sequential movements will be recorded and calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Fong-Chin Su, Principal Investigator — Chair Professor
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

REFERENCES:
- [Background] Organization, W.H., Global health and aging. Acedido março, 2011. 5: p. 2015.
- [Background] Grabiner MD, Enoka RM. Changes in movement capabilities with aging. Exerc Sport Sci Rev. 1995;23:65-104. No abstract available. PMID 7556361
- [Background] Ranganathan VK, Siemionow V, Sahgal V, Liu JZ, Yue GH. Skilled finger movement exercise improves hand function. J Gerontol A Biol Sci Med Sci. 2001 Aug;56(8):M518-22. doi: 10.1093/gerona/56.8.m518. PMID 11487606
- [Background] Olafsdottir HB, Zatsiorsky VM, Latash ML. The effects of strength training on finger strength and hand dexterity in healthy elderly individuals. J Appl Physiol (1985). 2008 Oct;105(4):1166-78. doi: 10.1152/japplphysiol.00054.2008. Epub 2008 Aug 7. PMID 18687981
- [Background] Keogh JW, Morrison S, Barrett R. Strength training improves the tri-digit finger-pinch force control of older adults. Arch Phys Med Rehabil. 2007 Aug;88(8):1055-63. doi: 10.1016/j.apmr.2007.05.014. PMID 17678670
- [Background] Kwok TC, Lam KC, Wong PS, Chau WW, Yuen KS, Ting KT, Chung EW, Li JC, Ho FK. Effectiveness of coordination exercise in improving cognitive function in older adults: a prospective study. Clin Interv Aging. 2011;6:261-7. doi: 10.2147/CIA.S19883. Epub 2011 Sep 29. PMID 22087065
- [Background] Zhang W, Scholz JP, Zatsiorsky VM, Latash ML. What do synergies do? Effects of secondary constraints on multidigit synergies in accurate force-production tasks. J Neurophysiol. 2008 Feb;99(2):500-13. doi: 10.1152/jn.01029.2007. Epub 2007 Nov 28. PMID 18046000
- [Background] Kim SW, Shim JK, Zatsiorsky VM, Latash ML. Finger inter-dependence: linking the kinetic and kinematic variables. Hum Mov Sci. 2008 Jun;27(3):408-22. doi: 10.1016/j.humov.2007.08.005. Epub 2008 Feb 5. PMID 18255182
- [Background] Shim JK, Lay BS, Zatsiorsky VM, Latash ML. Age-related changes in finger coordination in static prehension tasks. J Appl Physiol (1985). 2004 Jul;97(1):213-24. doi: 10.1152/japplphysiol.00045.2004. Epub 2004 Mar 5. PMID 15003998
- [Background] Parikh PJ, Cole KJ. Handling objects in old age: forces and moments acting on the object. J Appl Physiol (1985). 2012 Apr;112(7):1095-104. doi: 10.1152/japplphysiol.01385.2011. Epub 2012 Jan 12. PMID 22241054
- [Background] Shinohara M, Scholz JP, Zatsiorsky VM, Latash ML. Finger interaction during accurate multi-finger force production tasks in young and elderly persons. Exp Brain Res. 2004 Jun;156(3):282-92. doi: 10.1007/s00221-003-1786-9. Epub 2004 Feb 19. PMID 14985892
- [Background] Shinohara M, Li S, Kang N, Zatsiorsky VM, Latash ML. Effects of age and gender on finger coordination in MVC and submaximal force-matching tasks. J Appl Physiol (1985). 2003 Jan;94(1):259-70. doi: 10.1152/japplphysiol.00643.2002. Epub 2002 Sep 13. PMID 12391031
- [Background] Olafsdottir H, Zhang W, Zatsiorsky VM, Latash ML. Age-related changes in multifinger synergies in accurate moment of force production tasks. J Appl Physiol (1985). 2007 Apr;102(4):1490-501. doi: 10.1152/japplphysiol.00966.2006. Epub 2007 Jan 4. PMID 17204576
- [Background] Cobos, F.J.M. and M.d.M.M. Rodríguez, A Review of psychological intervention in Alzheimer s disease. International Journal of Psychology and Psychological Therapy, 2012. 12(3): p. 373-388.
- [Background] Franssen EH, Souren LE, Torossian CL, Reisberg B. Equilibrium and limb coordination in mild cognitive impairment and mild Alzheimer's disease. J Am Geriatr Soc. 1999 Apr;47(4):463-9. doi: 10.1111/j.1532-5415.1999.tb07240.x. PMID 10203123
- [Background] Verheij S, Muilwijk D, Pel JJ, van der Cammen TJ, Mattace-Raso FU, van der Steen J. Visuomotor impairment in early-stage Alzheimer's disease: changes in relative timing of eye and hand movements. J Alzheimers Dis. 2012;30(1):131-43. doi: 10.3233/JAD-2012-111883. PMID 22377783
- [Background] Wu YH, Pazin N, Zatsiorsky VM, Latash ML. Improving finger coordination in young and elderly persons. Exp Brain Res. 2013 Apr;226(2):273-83. doi: 10.1007/s00221-013-3433-4. Epub 2013 Feb 15. PMID 23411675
- [Background] Langlois F, Vu TT, Chasse K, Dupuis G, Kergoat MJ, Bherer L. Benefits of physical exercise training on cognition and quality of life in frail older adults. J Gerontol B Psychol Sci Soc Sci. 2013 May;68(3):400-4. doi: 10.1093/geronb/gbs069. Epub 2012 Aug 28. PMID 22929394
- [Background] Shim JK, Karol S, Kim YS, Seo NJ, Kim YH, Kim Y, Yoon BC. Tactile feedback plays a critical role in maximum finger force production. J Biomech. 2012 Feb 2;45(3):415-20. doi: 10.1016/j.jbiomech.2011.12.001. Epub 2012 Jan 4. PMID 22222494
- [Background] Kim Y, Shim JK, Hong YK, Lee SH, Yoon BC. Cutaneous sensory feedback plays a critical role in agonist-antagonist co-activation. Exp Brain Res. 2013 Aug;229(2):149-56. doi: 10.1007/s00221-013-3601-6. Epub 2013 Jul 9. PMID 23836110
- [Background] Li K, Marquardt TL, Li ZM. Removal of visual feedback lowers structural variability of inter-digit force coordination during sustained precision pinch. Neurosci Lett. 2013 Jun 17;545:1-5. doi: 10.1016/j.neulet.2013.04.011. Epub 2013 Apr 24. PMID 23624025
- [Background] Ambike S, Zatsiorsky VM, Latash ML. Processes underlying unintentional finger-force changes in the absence of visual feedback. Exp Brain Res. 2015 Mar;233(3):711-21. doi: 10.1007/s00221-014-4148-x. Epub 2014 Nov 23. PMID 25417192
- [Background] Hu X, Newell KM. Aging, visual information, and adaptation to task asymmetry in bimanual force coordination. J Appl Physiol (1985). 2011 Dec;111(6):1671-80. doi: 10.1152/japplphysiol.00760.2011. Epub 2011 Sep 29. PMID 21960656
- [Background] Seo NJ, Fischer HW, Bogey RA, Rymer WZ, Kamper DG. Use of visual force feedback to improve digit force direction during pinch grip in persons with stroke: a pilot study. Arch Phys Med Rehabil. 2011 Jan;92(1):24-30. doi: 10.1016/j.apmr.2010.08.016. Epub 2010 Nov 18. PMID 21092931
- [Background] Hu X, Loncharich M, Newell KM. Visual information interacts with neuromuscular factors in the coordination of bimanual isometric force. Exp Brain Res. 2011 Mar;209(1):129-38. doi: 10.1007/s00221-010-2528-4. Epub 2010 Dec 28. PMID 21188355
- [Background] Loucks TM, Ofori E, Sosnoff JJ. Force control under auditory feedback: effector differences and audiomotor memory. Percept Mot Skills. 2012 Jun;114(3):915-35. doi: 10.2466/24.25.27.PMS.114.3.915-935. PMID 22913030
- [Background] Jo HJ, Ambike S, Lewis MM, Huang X, Latash ML. Finger force changes in the absence of visual feedback in patients with Parkinson's disease. Clin Neurophysiol. 2016 Jan;127(1):684-692. doi: 10.1016/j.clinph.2015.05.023. Epub 2015 Jun 3. PMID 26072437
- [Background] Stein J, Bishop J, Gillen G, Helbok R. A pilot study of robotic-assisted exercise for hand weakness after stroke. IEEE Int Conf Rehabil Robot. 2011;2011:5975426. doi: 10.1109/ICORR.2011.5975426. PMID 22275627
- [Background] Wu YH, Truglio TS, Zatsiorsky VM, Latash ML. Learning to combine high variability with high precision: lack of transfer to a different task. J Mot Behav. 2015;47(2):153-65. doi: 10.1080/00222895.2014.961892. Epub 2014 Nov 3. PMID 25365477
- [Background] Friedman N, Chan V, Reinkensmeyer AN, Beroukhim A, Zambrano GJ, Bachman M, Reinkensmeyer DJ. Retraining and assessing hand movement after stroke using the MusicGlove: comparison with conventional hand therapy and isometric grip training. J Neuroeng Rehabil. 2014 Apr 30;11:76. doi: 10.1186/1743-0003-11-76. PMID 24885076
- [Background] Tsai, M.-F., 中風病人手指創新復健器. 成功大學生物醫學工程學系學位論文, 2016: p. 1-94.
- [Background] Levanon Y. The advantages and disadvantages of using high technology in hand rehabilitation. J Hand Ther. 2013 Apr-Jun;26(2):179-83. doi: 10.1016/j.jht.2013.02.002. PMID 23598084
- [Background] Manepalli, J., A. Desai, and P. Sharma, Psychosocial-environmental treatments for Alzheimer's disease. Primary Psychiatry, 2009. 16(6): p. 39.
- [Background] Chiu HY, Hsu HY, Kuo LC, Chang JH, Su FC. Functional sensibility assessment. Part I: develop a reliable apparatus to assess momentary pinch force control. J Orthop Res. 2009 Aug;27(8):1116-21. doi: 10.1002/jor.20859. PMID 19195027
- [Background] Hsu HY, Kuo LC, Chiu HY, Jou IM, Su FC. Functional sensibility assessment. Part II: Effects of sensory improvement on precise pinch force modulation after transverse carpal tunnel release. J Orthop Res. 2009 Nov;27(11):1534-9. doi: 10.1002/jor.20903. PMID 19402148
- [Background] Shieh SJ, Hsu HY, Kuo LC, Su FC, Chiu HY. Correlation of digital sensibility and precision of pinch force modulation in patients with nerve repair. J Orthop Res. 2011 Aug;29(8):1210-5. doi: 10.1002/jor.21365. Epub 2011 Mar 4. PMID 21374708
- [Background] Hsu HY, Kuo LC, Kuo YL, Chiu HY, Jou IM, Wu PT, Su FC. Feasibility of a novel functional sensibility test as an assisted examination for determining precision pinch performance in patients with carpal tunnel syndrome. PLoS One. 2013 Aug 20;8(8):e72064. doi: 10.1371/journal.pone.0072064. eCollection 2013. PMID 23977209
- [Background] Yen WJ, Kuo YL, Kuo LC, Chen SM, Kuan TS, Hsu HY. Precision pinch performance in patients with sensory deficits of the median nerve at the carpal tunnel. Motor Control. 2014 Jan;18(1):29-43. doi: 10.1123/mc.2013-0004. PMID 24496877
- [Background] Chiu HY, Hsu HY, Su FC, Jou IM, Lin CF, Kuo LC. Setup of a novel biofeedback prototype for sensorimotor control of the hand and preliminary application in patients with peripheral nerve injuries. Phys Ther. 2013 Feb;93(2):168-78. doi: 10.2522/ptj.20120050. Epub 2012 Sep 27. PMID 23023814
- [Background] Hsu HY, Lin CF, Su FC, Kuo HT, Chiu HY, Kuo LC. Clinical application of computerized evaluation and re-education biofeedback prototype for sensorimotor control of the hand in stroke patients. J Neuroeng Rehabil. 2012 May 9;9:26. doi: 10.1186/1743-0003-9-26. PMID 22571177
- [Background] Hsu HY, Kuo LC, Jou IM, Chen SM, Chiu HY, Su FC. Establishment of a proper manual tactile test for hands with sensory deficits. Arch Phys Med Rehabil. 2013 Mar;94(3):451-8. doi: 10.1016/j.apmr.2012.07.024. Epub 2012 Aug 9. PMID 22885285
- [Background] Hsu HY, Kuo YL, Jou IM, Su FC, Chiu HY, Kuo LC. Diagnosis from functional perspectives: usefulness of a manual tactile test for predicting precision pinch performance and disease severity in subjects with carpal tunnel syndrome. Arch Phys Med Rehabil. 2014 Apr;95(4):717-25. doi: 10.1016/j.apmr.2013.11.017. Epub 2013 Dec 16. PMID 24355426
- [Background] Hsu HY, Shieh SJ, Kuan TS, Yang HC, Su FC, Chiu HY, Kuo LC. Manual Tactile Test Predicts Sensorimotor Control Capability of Hands for Patients With Peripheral Nerve Injury. Arch Phys Med Rehabil. 2016 Jun;97(6):983-90. doi: 10.1016/j.apmr.2016.01.008. Epub 2016 Jan 30. PMID 26829761
- [Background] Chiu HY, Hsu HY, Kuo LC, Su FC, Yu HI, Hua SC, Lu CH. How the impact of median neuropathy on sensorimotor control capability of hands for diabetes: an achievable assessment from functional perspectives. PLoS One. 2014 Apr 10;9(4):e94452. doi: 10.1371/journal.pone.0094452. eCollection 2014. PMID 24722361
- [Background] Hsu HY, Chiu HY, Lin HT, Su FC, Lu CH, Kuo LC. Impacts of elevated glycaemic haemoglobin and disease duration on the sensorimotor control of hands in diabetes patients. Diabetes Metab Res Rev. 2015 May;31(4):385-94. doi: 10.1002/dmrr.2623. Epub 2015 Feb 3. PMID 25417846
- [Background] Yang CJ, Hsu HY, Lu CH, Chao YL, Chiu HY, Kuo LC. The associations among hand dexterity, functional performance, and quality of life in diabetic patients with neuropathic hand from objective- and patient-perceived measurements. Qual Life Res. 2015 Jan;24(1):213-21. doi: 10.1007/s11136-014-0748-y. Epub 2014 Jul 14. PMID 25017499
- [Background] Chen PT, Jou IM, Lin CJ, Chieh HF, Kuo LC, Su FC. Is the Control of Applied Digital Forces During Natural Five-digit Grasping Affected by Carpal Tunnel Syndrome? Clin Orthop Relat Res. 2015 Jul;473(7):2371-82. doi: 10.1007/s11999-015-4189-x. Epub 2015 Feb 18. PMID 25690168
- [Background] Chen PT, Lin CJ, Jou IM, Chieh HF, Su FC, Kuo LC. One digit interruption: the altered force patterns during functionally cylindrical grasping tasks in patients with trigger digits. PLoS One. 2013 Dec 31;8(12):e83632. doi: 10.1371/journal.pone.0083632. eCollection 2013. PMID 24391799
- [Background] Kuo LC, Chen SW, Lin CJ, Lin WJ, Lin SC, Su FC. The force synergy of human digits in static and dynamic cylindrical grasps. PLoS One. 2013;8(3):e60509. doi: 10.1371/journal.pone.0060509. Epub 2013 Mar 27. PMID 23544151
- [Background] Kuo LC, Hsu HM, Wu PT, Lin SC, Hsu HY, Jou IM. Impact of distal median neuropathy on handwriting performance for patients with carpal tunnel syndrome in office and administrative support occupations. J Occup Rehabil. 2014 Jun;24(2):332-43. doi: 10.1007/s10926-013-9471-8. PMID 23934582
- [Background] Hsu, H.-M., et al., Quantification of handwriting performance: Development of a force acquisition pen for measuring hand-grip and pen tip forces. Measurement, 2013. 46(1): p. 506-513.
- [Background] Lai, K.-Y., et al., Effects of hand span size and right-left hand side on the piano playing performances: Exploration of the potential risk factors with regard to piano-related musculoskeletal disorders. International Journal of Industrial Ergonomics, 2015. 50: p. 97-104.
- [Background] Park J, Wu YH, Lewis MM, Huang X, Latash ML. Changes in multifinger interaction and coordination in Parkinson's disease. J Neurophysiol. 2012 Aug 1;108(3):915-24. doi: 10.1152/jn.00043.2012. Epub 2012 May 2. PMID 22552184